CLINICAL TRIAL: NCT02010749
Title: Protein Concentration in Infant Formula: A Follow-up Study of Growth at 2 Years of Age
Status: Completed | Type: Observational
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Other Study IDs: 9052A1-3001 PHL
Record Dates: First submitted 2013-11-06; First posted 2013-12-13 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-12

CONDITIONS: Bottle Feeding
MeSH Terms: conditions — Bottle Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — stool
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control: Control: Children who had received Standard formula (SF) as infants
- Experimental: Experimental: Children who had received lower protein formula as infants

SUMMARY:
The primary objective of the study was to compare the growth parameters of children approximately 2* years of age, who as infants were randomized to receive either a lower-protein formula ("experimental formula"; EF) with 12.8 g/L protein or a standard formula (SF) with 14.1 g/L protein or who were human milk (HM) fed for the first 4 months of life. The secondary objective was to describe diet and nutrient intake in this cohort of children. The exploratory objectives were to describe stool microbiota in a subset of this cohort and stool composition (stool soap and nonsoap fatty acids, total fatty acids, and minerals) in a second subset of this cohort.

(* The mean age of subjects was 33.0 months due to a delay in the study start-up.)

DETAILED DESCRIPTION:
This was an observational, single-site, follow-up study of healthy children who as infants who had completed study 9052A1-3000. An attempt was made to contact all subjects who had completed study 9052A1-3000 by telephone to ask them to participate in study 9052A1-3001. Approximately 66 and 60 subjects were planned to participate in the stool microbiota and stool composition substudies, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Children who were enrolled in the Wyeth Nutrition study are eligible to participate in this study

Exclusion Criteria:

* Children who were not enrolled in the Wyeth Nutrition study are not eligible to participate in this study
* Children who have received any antibiotics and antifungal medications except topical within two weeks prior to enrollment are not eligible to participate in the stool microbiota study
* Children who are taking any medications known or suspected to affect fat digestion, absorption, and or metabolism, any vitamin and or mineral supplements which contain calcium, suppositories, bismuth-containing medications, herbal supplements, or medications that may neutralize or suppress gastric acid secretion, are not eligible to participate in the stool composition study

Ages: 2 Years to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children 2 years of age who were enrolled in the Wyeth Nutrition study
Sampling Method: Probability Sample
Enrollment: 267 (Actual)
Dates: Start 2010-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Weight-for-Length Z-Scores | 2 years of age
  Primary Efficacy Endpoint: weight-for-length Z-score based on World Health Organization (WHO) growth charts.

SECONDARY OUTCOMES:
Weight-for-age Z-score | 2 years of age
  Weight-for-age Z-score based on World Health Organization (WHO) growth charts
Length-for-age Z-score | 2 years of age
  Length-for-age Z-score based on World Health Organization (WHO) growth charts
Head circumference-for-age Z-score | 2 years of age
  Head circumference-for-age Z-score based on World Health Organization (WHO) growth charts
BMI-for-age Z-score | 2 years of age
  BMI-for-age Z-score based on WHO and Centers for Disease Control (CDC) growth charts
Dietary intake | 2 years of age
  Dietary intake (servings per day), percent contribution to energy intake, and percent contribution to protein intake of Dietary endpoints included mean intake (servings per day), percentage contribution to energy intake, and percentage contribution to protein intake of:
  * Cereal/cereal products
  * Starchy roots/tubers
  * Sugars/syrups
  * Fats/oils
  * Fish/meat/poultry
  * Eggs
  * Milk and milk products
  * Dried beans/nuts/seeds
  * Vegetables
  * Fruits
  * Miscellaneous foods
Nutrient intake | 2 years of age
  Nutrition endpoints included mean intake and percentage adequacy based on the recommended intake of:
  * Total energy (kcal)
  * Protein (g)
  * Carbohydrates (g) (mean intake only)
  * Fat (g) (mean intake only)
  * Iron (mg)
  * Retinol equivalents (μg)
  * Calcium (g)
  * Thiamin (mg)
  * Riboflavin (mg)
  * Niacin (mg)
  * Ascorbic acid (mg)
  * Iodine (μg)
  * Vitamin D (μg)
  * Zinc (μg)

OTHER OUTCOMES:
Stool microbiota Follow-up Study of Growth at 2 Years of Age | 2 years of age
  Stool microbiota included relative abundance of the following classes of bacteria, expressed as a percentage of total bacteria:
  * Bifidobacteria
  * Bacteroides
  * Clostridia
  * Enterobacteriaceae
  * Lactobacilli
  * Streptococci
Stool composition | 2 years of age
  quantitative measures of the following parameters in stool wet and dry weight:
  * Total soap fatty acids (%)
  * Individual soap fatty acids (C12:0, C14:0, C16:0, C18:0, C18:1, C18:2) (mg/g)
  * Nonsoap fatty acids (%)
  * Total fatty acids (%)
  * Total lipids (%)
  * Soap lipids (%)
  * Nonsoap lipids (%)
  * Minerals: calcium (%), magnesium (%), and phosphorus (%)
  * Nitrogen (%) In addition, stool solids and stool moisture were assessed as percentage of stool wet weight only.
Incidence of adverse events | 2 years of age
  Safety was evaluated from signing of the informed consent to study completion, through the recording and monitoring of adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Asian Hospital and Medical Center, Filinvest Corporate City, Alabang,, Muntinlupa City, Philippines

REFERENCES:
- [Derived] Gonzalez-Garay AG, Serralde-Zuniga AE, Medina Vera I, Velasco Hidalgo L, Alonso Ocana MV. Higher versus lower protein intake in formula-fed term infants. Cochrane Database Syst Rev. 2023 Nov 6;11(11):CD013758. doi: 10.1002/14651858.CD013758.pub2. PMID 37929831